CLINICAL TRIAL: NCT02951520
Title: A Novel Single-puncture Triple Nerve Block; Sciatic, Obturator, Femoral Technique (SOFT), as a Sole Anesthesia for Knee Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Healthpoint Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Muhammad Taha, Consultant of anesthesia, Healthpoint Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC 001
Record Dates: First submitted 2016-10-29; First posted 2016-11-01 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Arthroscopic Knee Ligament Reconstruction
Keywords: Patients

ARMS (1):
- SOFT block (Experimental): Fifty patients will form the study group (one group). All the patients will receive supine ultrasound guided (US) sciatic, obturator, femoral nerve block technique using a single skin puncture (SOFT block).
  Interventions: Procedure: new technique for lower limb nerve blocks using a single skin puncture (SOFT block)

INTERVENTIONS:
Procedure: new technique for lower limb nerve blocks using a single skin puncture (SOFT block) — The patients will be in supine position. The block needle will be inserted at the inguinal crease (medial to the femoral vein) and advanced towards the femoral nerve, then redirected towards the obturator nerve (deep to the pectineus muscle). Lastly, it will be redirected posteriorly towards the sciatic nerve (deep to the quadratus femoris muscle). A ropivacaine-lidocaine-epinephrine mixture will be used to block these nerves. The block success rate (painless surgery), performance time and patient discomfort will be recorded.

SUMMARY:
This study aims to describe and to evaluate the effectiveness (success rate) of a supine ultrasound (US) guided single-puncture sciatic, obturator and femoral neve block technique (SOFT block) in knee surgery.

DETAILED DESCRIPTION:
Under aseptic technique, all the patients will receive US-guided femoral, obturator and sciatic nerve blocks using a single puncture point. All blocks will be performed by an expert anesthetist. The femoral nerve will be blocked lateral to the femoral artery. The obturator nerve will be blocked after it exits the obturator canal (deep to pectineus muscle). While the sciatic nerve will be blocked deep (posterior) to the inferior border of quadratus femoris muscle. The motor block of the femoral, obturator and sciatic nerves and sensory block of the lateral femoral cutaneous nerve (LFCN) will be assessed before shifting the patient to the operating room.

The performance time, patient discomfort, technique success rate, the associated successful LFCN block and any complication will be recorded by the assistant. All patients were assessed neurologically before discharge and during the physiotherapy visits for 3 weak after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for arthroscopic knee ligament reconstruction

Exclusion Criteria:

* BMI > 30 kg.m-2,
* ASA physical state >II
* Allergy to the used local anesthetics
* Infection at the injection site
* age <18y

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
success rate | within the perioperative period

CONTACTS AND LOCATIONS:
Locations (1):
- Healthpoint Hospital, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates